CLINICAL TRIAL: NCT00871832
Title: To Evaluate if Pre-admission Hyperglycemia Measured by Glycosylated Hemoglobin Level Affects the Morbidity and Mortality of Patients in a Mixed Medical and Surgical Intensive Care Unit
Brief Title: Pre-admission Hyperglycemia and Its Effect on Morbidity and Mortality
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Mario Castellanos, Clinical Director of Research, Dept. of Medicine, Northwell Health
Other Study IDs: 07-020
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Hyperglycemia
Keywords: hyperglycemia; HgA1c; mortality
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is currently standard of care in many Medical and Surgical ICU's to institute a nurse driven insulin protocol in maintaining tight glucose control in the critical patient. Many articles have been written to address this topic. However, there is no current data regarding the use of glycohemoglobin as a marker of risk of morbidity and mortality. In our study we would like to determine whether or not the HbA1C could be used as a marker of morbidity and mortality. The HbA1C is a simple blood test that may be added on to any CBC collection tube; a blood sample that critical patients have drawn up to several times a day. The investigators would analyze this information in respect to the rest of the clinical data collected regarding the patient's illness.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the medical and surgical ICU, and CCU that are 18 year's or older and speak English that give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the medical and surgical ICU, and CCU that are 18 year's or older and speak English that give consent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
morbidity and mortality | at time of review
  looking to see if HbA1C correlates with morbidity (i.e. sepsis, renal failure, length of stay) or death

CONTACTS AND LOCATIONS:
Overall Officials: Mario Castellanos, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States